CLINICAL TRIAL: NCT03178331
Title: Who Benefit From School Doctors' Health Checks: a Prospective Study of a Screening Method in Finland
Brief Title: Who Benefit From School Doctors' Health Checks?
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Päivikki and Sakari Sohlberg Foundation, Finland (Other); City of Helsinki (Other); Finnish Foundation for General Practice (Unknown); General Practitioners in Finland (Unknown); Network of Academic Health Centres, Finland (Unknown); Foundation for Paediatric Research, Finland (Other); Pediatric Research Center, University of Helsinki (Unknown)
Responsible Party: Principal Investigator, Kirsi Nikander, Principal Investigator, University of Helsinki
Other Study IDs: HUS/2174/2017
Record Dates: First submitted 2017-05-29; First posted 2017-06-06 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: School Health Services
Keywords: Children; Student; Questionnaires; Screening; Health check; School health services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grade 1 children: Areas of concern in study questionnaires: growth, physical symptom, hearing, school absenteeism, learning, concentration, behavior, emotions, getting on with others, eating, sleeping, wellbeing of family, free description of concern, wish to talk about concerns with the school doctor
  Interventions: Other: Study questionnaires
- Grade 5 children: Areas of concern in study questionnaires: growth, physical symptom, hearing, school absenteeism, learning, concentration, behavior, emotions, getting on with others, eating, sleeping, wellbeing of family, free description of concern, wish to talk about concerns with the school doctor
  Interventions: Other: Study questionnaires

INTERVENTIONS:
Other: Study questionnaires — filled by parents, school nurse and teacher

SUMMARY:
The aims of the study are 1) to evaluate the potential benefits or harm of school doctors' routine health checks and 2) to explore whether part of the school doctors' routine health checks can be omitted using study questionnaires which address the parents', school nurses' and teachers' concerns regarding each child.

DETAILED DESCRIPTION:
The aim is to include 4 cities, 21 schools, 14 doctors and 1050 children from Southern Finland. From each doctor the aim is to get 25 children from both grades 1 and 5 (at ages 7 and 11) from 1-2 schools. Before the school doctor's check-up, the parents, nurses and teachers fill a questionnaire to identify any potential concerns about each child. The questions were partly chosen from the Strengths and Difficulties Questionnaire (SDQ). Additional questions concerning the child's growth, physical well-being, learning, school absenteeism and the well-being of the whole family are included. The doctor is blinded to the answers of the questionnaires. After the health check the doctors fill an electronic report including any instructions given, significant discussions and follow-up plans and their estimate of the potential benefit or harm of the medical appointment. The child and the parent fill patient-reported experience measure (PREM) forms where they evaluate the benefit or harm of the health check. The researchers compare the need for a doctor's appointment to the benefit gained. At one year after the check-up, the implementations of the follow-up plans are analyzed.

A data balance sheet has been prepared. The coordinating ethics committee of the Hospital District of Helsinki and Uusimaa (HUS) has approved the study protocol. Permissions for the study from the Department of Social Services and Healthcare and the Department of Education from all participating cities have been obtained. Informed consent will be obtained from all participating children, parents, doctors, nurses and teachers.

ELIGIBILITY:
Inclusion Criteria:

Grade 1 and grade 5 children

Exclusion Criteria:

Children studying mainly in special education groups or the need of an interpreter

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Finnish public primary schools from four urban municipalities (Helsinki, Tampere, Kirkkonummi and Kerava) in Southern Finland
Sampling Method: Probability Sample
Enrollment: 1013 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
The need for a school doctor's health check | Baseline
  The need for a school doctor's health check according to the study questionnaires filled by parents, nurse and teacher.
  Areas of concern in study questionnaires: growth, physical symptom, hearing, school absenteeism, learning, concentration, behavior, emotions, getting on with others, eating, sleeping, wellbeing of family, free description of concern, wish to talk about concerns with the school doctor
  The responses will be categorized into three groups: 1) "Needs doctor's health check" 2) "No need for doctor's health check and 3) "Consultation of the nurse or doctor may be sufficient".
The benefit/harm of school doctors' routine health checks | Baseline
  A seven point likert scale that is based on:
  1. Measures from the doctor's electronic report: instruction, other significant discussion, referral to laboratory test/physiotherapist/speech therapist/nutritionist/secondary care, guidance to or contact of a specialised worker or other unit: teacher/special education teacher/school psychologist/school social worker/health center/family guidance center/home service/child welfare, prescription, medical imaging, individual follow-up plan
  2. School doctor's evaluation of benefit/harm
  3. Patient reported experience measures (PREM) of benefit/harm by child and parent

SECONDARY OUTCOMES:
Interventions and plans arising from school doctors' routine health checks | Baseline
  Measures from the doctor's electronic report: instruction, other significant discussion, referral to laboratory test/physiotherapist/speech therapist/nutritionist/secondary care, guidance to or contact of a specialised worker or other unit: teacher/special education teacher/school psychologist/school social worker/health center/family guidance center/home service/child welfare, prescription, medical imaging, individual follow-up plan
The implementations of the school doctors' follow-up plans | 12 months
  The implementations of measures from the doctor's electronic report (yes, no, information not accessible): instruction, referral to laboratory test/physiotherapist/speech therapist/nutritionist/secondary care, guidance to or contact of a specialised worker or other unit: teacher/special education teacher/school psychologist/school social worker/health center/family guidance center/home service/child welfare, prescription, medical imaging, individual follow-up plan

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi M Nikander, MD, PhD, Principal Investigator — Doctoral School in Health Sciences, University of Helsinki, Finland; Elina Hermanson, MD, PhD, Study Director — Pikkujätti Medical Centre for Children and Youth, Finland; Silja Kosola, MD, PhD, Study Director — Helsinki University Hospital and University of Helsinki, Finland; Minna Kaila, Professor, Study Chair — Faculty of Medicine, University of Helsinki, Finland
Locations (4):
- Finland (4):
  - School and Student Health Services, Helsinki
  - School and Student Health Services, Kerava
  - School and Student Health Services, Kirkkonummi
  - School and Student Health Services, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nikander K, Hermanson E, Vahlberg T, Kaila M, Kosola S. Parent, teacher, and nurse concerns and school doctor actions: an observational study of general health checks. BMJ Open. 2022 Nov 15;12(11):e064699. doi: 10.1136/bmjopen-2022-064699. PMID 36379665
- [Derived] Nikander K, Kosola S, Vahlberg T, Kaila M, Hermanson E. Associating school doctor interventions with the benefit of the health check: an observational study. BMJ Paediatr Open. 2022 Feb;6(1):e001394. doi: 10.1136/bmjpo-2021-001394. PMID 36053658
- [Derived] Nikander K, Hermanson E, Vahlberg T, Kaila M, Sannisto T, Kosola S. Associations between study questionnaire-assessed need and school doctor-evaluated benefit of routine health checks: an observational study. BMC Pediatr. 2021 Aug 16;21(1):346. doi: 10.1186/s12887-021-02810-0. PMID 34399731
- [Derived] Nikander K, Kosola S, Kaila M, Hermanson E. Who benefit from school doctors' health checks: a prospective study of a screening method. BMC Health Serv Res. 2018 Jun 27;18(1):501. doi: 10.1186/s12913-018-3295-3. PMID 29945604